CLINICAL TRIAL: NCT00249015
Title: Randomized Controlled Trial of Combined Aerobic and Resistance Exercise in Breast Cancer Survivors. The CARE Trial.
Brief Title: Trial of Combined Aerobic and Resistance Exercise in Breast Cancer Survivors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: BR-01-0080 ethics 22148
Record Dates: First submitted 2005-11-04; First posted 2005-11-07 (Estimated); Last update posted 2016-07-18 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: aerobic exercise; resistance exercise; physical fitness; body composition; quality of life; rehabilitation; psychosocial oncology; adherence
MeSH Terms: conditions — Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Combined Aerobic and Resistance Exercise Program: perform three exercise sessions per week consisting of about 25-30 minutes of aerobic exercise at a moderate-to-vigorous intensity as well as some weight training consisting of two sets of 8-12 repetitions of 9-10 different exercises. For the aerobic exercise, participant can choose from different exercise equipment such as a treadmill or stationary bicycle.
  Interventions: Behavioral: Physical exercise
- 2 (Active Comparator): Moderate Aerobic Exercise Group: perform three exercise sessions per week consisting of about 25-30 minutes of aerobic exercise at a moderate-to-vigorous intensity. Again, participant can choose from different exercise equipment.
  Interventions: Behavioral: Physical exercise
- 3 (Experimental): High Aerobic Exercise Group: perform three exercise sessions per week consisting of about 45-60 minutes of aerobic exercise at a moderate-to-vigorous intensity. Again, participant can choose from different exercise equipment.
  Interventions: Behavioral: Physical exercise

INTERVENTIONS:
Behavioral: Physical exercise — perform exercise program 3 days per week and 5 minutes of warm-up and cool-down exercises before and after the main exercise component

SUMMARY:
Endurance exercise such as walking has been shown to help breast cancer survivors maintain their energy and quality of life while they are receiving chemotherapy, but there have not been any studies on weight training. In this study, the researchers want to determine if a combined program of endurance and weight training exercises is better than a standard amount of endurance exercise or even a higher amount of endurance exercise in breast cancer survivors receiving chemotherapy. The study will be an experimental design in which the researchers have breast cancer survivors participate in one of the three different exercise programs. The researchers' main interest is in patient rated physical functioning and quality of life, which they will measure before and after the exercise programs by asking participants how they feel on various rating scales. The researchers will also measure their aerobic fitness on a treadmill and how strong they are by having them lift weights.

DETAILED DESCRIPTION:
BACKGROUND: Aerobic exercise has been shown to improve physical fitness and quality of life (QoL) in breast cancer survivors receiving chemotherapy but no study to date has examined the addition of resistance exercise to aerobic exercise in this population. Resistance exercise has proven to be an important adjunct to aerobic exercise in the cardiac rehabilitation population although few trials have controlled for the total volume of exercise.

PURPOSE: The primary purpose of the present trial is to compare the effects of a combined aerobic and resistance exercise program (COMB) to a standard moderate volume of aerobic exercise (STAN) and a higher volume of aerobic exercise (HIGH) that controls for the total volume of exercise in the COMB arm.

METHODS: The study will be a prospective, three-armed, randomized controlled trial conducted in Edmonton (coordinating center), Ottawa, and Vancouver. Participants will be 300 breast cancer survivors scheduled to receive adjuvant chemotherapy. All three exercise groups will be asked to perform supervised exercise 3 days/week for the length of their chemotherapy treatment. The STAN group will be asked to perform approximately 500 kilocalories/week of self-selected aerobic activities (e.g., treadmill, cycle ergometer, elliptical). This arm of the trial is considered standard care based on the emerging consensus of recent systematic reviews and recommendations from major cancer agencies. The HIGH group will be asked to complete approximately 1,000 kilocalories/week of self-selected aerobic activities. The COMB group will be asked to complete 1,000 kilocalories/week split equally between aerobic and resistance exercise. The primary endpoint in the trial will be change in physical functioning between baseline and post intervention as assessed by the physical functioning subscale of the Short Form (SF) 36 scale. Secondary endpoints will include cardiorespiratory fitness (maximal treadmill test), muscular strength (8 repetition maximum tests), muscular endurance (standard load test at 50% of estimated baseline maximum), body composition (DEXA scans), psychological distress, sleep quality, exercise adherence, and chemotherapy completion rates.

RELEVANCE: An important issue for breast cancer survivors receiving chemotherapy is whether there is any advantage to increasing the volume of aerobic exercise or adding resistance exercise to a standard aerobic exercise program. If there is an advantage, then it is important that breast cancer survivors receive this optimal exercise prescription to maximize their ability to cope with their chemotherapy treatments and maintain their physical function and QoL during this difficult time.

ELIGIBILITY:
* Are diagnosed with stage I-IIIA breast cancer, histologically confirmed
* Are scheduled to receive adjuvant chemotherapy (receiving neoadjuvant chemotherapy for locally advanced cancer is an exclusion criteria)
* Have not received previous chemotherapy (previous cancer is NOT an exclusion criteria)
* Have not received transabdominal rectus abdominis muscle (TRAM) reconstructive surgery
* Are 18 years or older
* Received approval from their treating oncologist
* No uncontrolled hypertension, cardiac illness or psychiatric condition or any other medical condition that would be a contraindication to exercise
* Able to understand and provide written informed consent in English or French (Ottawa)
* Complete maximal aerobic and strength tests. No contraindication to exercise as determined by fitness tests
* Are not pregnant
* Willing to accept randomization and complete their assigned exercise program
* If participant is currently exercising (e.g., swimming at the Y 3 times per week) must be willing to give this up in place of their randomly assigned program
* Willing to travel to fitness center 3 times/week to complete exercise program
* Willing to complete all assessments (except blood) at all timepoints including 6, 12, and 24 month follow-ups
* Must not have a planned/known absence of greater than 2 weeks during the intended intervention period and must be able/willing to perform exercise sessions on their own during any planned absences of less than 2 weeks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2008-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Patient rated physical functioning | at 8 weeks and 24 weeks

SECONDARY OUTCOMES:
Physical fitness, body composition, treatment completion rates, exercise adherence rates, adverse events | at 8 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kerry Courneya, PhD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada

REFERENCES:
- [Derived] An KY, Arthuso FZ, Kang DW, Morielli AR, Ntoukas SM, Friedenreich CM, McKenzie DC, Gelmon K, Mackey JR, Courneya KS. Exercise and health-related fitness predictors of chemotherapy completion in breast cancer patients: pooled analysis of two multicenter trials. Breast Cancer Res Treat. 2021 Jul;188(2):399-407. doi: 10.1007/s10549-021-06205-8. Epub 2021 Mar 29. PMID 33779887
- [Derived] An KY, Kang DW, Morielli AR, Friedenreich CM, Reid RD, McKenzie DC, Gelmon K, Mackey JR, Courneya KS. Patterns and predictors of exercise behavior during 24 months of follow-up after a supervised exercise program during breast cancer chemotherapy. Int J Behav Nutr Phys Act. 2020 Feb 14;17(1):23. doi: 10.1186/s12966-020-00924-9. PMID 32059728
- [Derived] Courneya KS, Segal RJ, Vallerand JR, Forbes CC, Crawford JJ, Dolan LB, Friedenreich CM, Reid RD, Gelmon K, Mackey JR, McKenzie DC. Motivation for Different Types and Doses of Exercise During Breast Cancer Chemotherapy: a Randomized Controlled Trial. Ann Behav Med. 2016 Aug;50(4):554-63. doi: 10.1007/s12160-016-9782-z. PMID 26896305